CLINICAL TRIAL: NCT02228044
Title: Alcohol, Suicide, and HIV Prevention for Teens in Mental Health Treatment
Brief Title: Alcohol, Suicide and HIV Prevention for Teens in Mental Health Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5970; R01AA016854 (NIH)
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Suicide; Alcohol Abuse; Drug Abuse; HIV
Keywords: suicide; alcohol; marijuana; HIV; prevention; adolescent
MeSH Terms: conditions — Suicide; Alcoholism; Substance-Related Disorders; Marijuana Abuse | interventions — National Program of Cancer Registries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prevention Program (Experimental): This is a cognitive-behavioral substance abuse, suicide, and HIV prevention program delivered in a workshop format to adolescent participants and their parents/legal guardians.
  Interventions: Behavioral: Prevention program
- Assessment Only (No Intervention)

INTERVENTIONS:
Behavioral: Prevention program
  Arms: Prevention Program

SUMMARY:
This study examines whether an integrated alcohol/substance abuse, suicide, and HIV prevention protocol is associated with lower onset and frequency of alcohol and other drug use, suicidal behavior, and high risk sexual behavior among adolescents receiving community based mental health care.

DETAILED DESCRIPTION:
The purpose of this study is to compare an integrated adolescent alcohol/drug, suicide, and HIV prevention program to an assessment only control condition in a randomized clinical trial. This prevention protocol is designed as an "add-on" intervention to standard mental health care. We will examine the extent to which the addition of this prevention protocol is associated with lower rates of alcohol use and drug use, suicidal behavior, and HIV related risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* ages 13-18
* English speaking adolescent and at least one English speaking parent
* receiving mental health treatment
* living with a parent or guardian willing to participate

Exclusion Criteria:

* Active Alcohol or Marijuana Dependence Diagnosis
* HIV infection
* Pregnant
* Current psychosis
* Cognitively unable to give assent

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2008-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
adolescent alcohol use and binge drinking (any, number of days, number of related problems) | change from baseline to 6 months (prior 3 months)
  This was assessed using the Customary Drinking and Drug Use Record
adolescent suicidal ideation and behavior (severity of suicidal ideation and presence of any suicidal ideation or suicidal behavior) | change from baseline to 6 months (prior month to 6 months)
  This was assessed using the Suicidal ideation Questionnaire and the Self-Injurious Thoughts and Behavior Interview
adolescent HIV risk behavior (any sexual behavior, number of sexual partners, number of unprotected sexual acts) | change from baseline to 6 months (prior 3 months)
  This was assessed using the Adolescent Risk Behavior Assessment.
adolescent marijuana use (any use, number of days, related problems) | change from baseline to 6 months (prior 3 months)
  This was assessed with the Customary Drinking and Drug Use Measure
adolescent alcohol use and binge drinking (any, number of days, number of related problems) | change from baseline to 12 months (prior 3 months)
  This was assessed using the Customary Drinking and Drug Use Measure
adolescent suicidal ideation and behavior (severity of suicidal ideation and presence of any suicidal ideation or suicidal behavior) | change from baseline to 12 months (prior month to 6 months)
  This was assessed with the Suicidal Ideation Questionnaire and the Self-Injurious Thoughts and Behavior Questionnaire
adolescent HIV risk behavior (any sexual behavior, number of sexual partners, number of unprotected sexual acts) | change from baseline to 12 months (prior 3 months)
  This was assessed with the Adolescent Risk Behavior Assessment
adolescent marijuana use (any use, number of days, related problems) | change from baseline to 12 months (prior 3 months)
  This was assessed with the Customary Drinking and Drug Use Record

SECONDARY OUTCOMES:
frequency of parental monitoring behavior | change from baseline to 1 month
  This was assessed with the Parental Monitoring Questionnaire
quality of parent-child communication around high risk behaviors | change from baseline to 1 month
  This was assessed with the Parent-Adolescent Sexual Communication Scale and items adapted for alcohol/drug use and suicidal behavior
adolescent perceptions of parental degree of disapproval of high risk behavior | change from baseline to 1 month
  This was assessed with Parental Norms for Sexual Activity and Supervision Scale and items adapted for alcohol/drug use
adolescent perception of degree of interpersonal coping and stress management skills | change from baseline to 6 months
  This was assessed with the Bar-On Emotional Quotient Inventory - Youth Version
adolescent degree of perceived self-efficacy for condom use | change from baseline to 1 month
  This was assessed with the Self-Efficacy for Condom Use Scale
adolescent degree of HIV related knowledge | change from baseline to 1 month
  This was assessed with the HIV Knowledge Scale
adolescent perceptions of degree of peer substance use and tolerance of use | change from baseline to 6 months
  This was assessed with Peer Substance Use and Tolerance of Use scale
adolescent perception of the degree of peer approval of sexual activity | change from baseline to 6 months
  This was assessed with the Peer Norms Scale for Sexual Activity scale
adolescent degree of perceived self-efficacy for HIV prevention | change from baseline to 1 month
  This was assessed with the Self-Efficacy for HIV Prevention Scale
frequency of positive and negative thoughts related to suicide | change from baseline to 1 month
  This was assessed with the Positive and Negative Suicide Ideation Inventory
degree of adolescent positive/negative attitudes and beliefs about alcohol | change from baseline to 1 month
  This was assessed with the Youth Alcohol and Drug Survey
degree of adolescent positive/negative attitudes and beliefs about marijuana use | change from baseline to 1 month
  This was assessed with the Youth Alcohol and Drug Survey
frequency of parental monitoring behavior | change from baseline to 6 months
  This was assessed with the parental monitoring questionnaire
frequency of parental monitoring behavior | change from baseline to 12 months
  This was assessed with the parental monitoring questionnaire
quality of parent-child communication around high risk behaviors | change from baseline to 6 months
  This was assessed with the Parent-Adolescent Sexual Communication Scale and items adapted for alcohol/drug use and suicidal behavior
quality of parent-child communication around high risk behaviors | change from baseline to 12 months
  This was assessed with the Parent-Adolescent Sexual Communication Scale and items adapted for alcohol/drug use and suicidal behavior
adolescent perceptions of parental degree of disapproval of high risk behavior | change from baseline to 6 months
  This was assessed with Parental Norms for Sexual Activity and Supervision Scale and items adapted for alcohol/drug use
adolescent perceptions of parental degree of disapproval of high risk behavior | change from baseline to 12 months
  This was assessed with Parental Norms for Sexual Activity and Supervision Scale and items adapted for alcohol/drug use
adolescent perception of degree of interpersonal and stress management coping skills | change from baseline to 12 months
  This was assessed with the Bar-On Emotional Quotient Inventory - Youth Version
adolescent perceptions of degree of peer substance use and approval of use | change from baseline to 12 months
  This was assessed with Peer Substance Use and Tolerance of Use scale
adolescent perception of the degree of peer approval of sexual activity | change from baseline to 12 months
  This was assessed with the Peer Norms Scale for Sexual Activity scale

CONTACTS AND LOCATIONS:
Overall Officials: Christianne Esposito-Smythers, Ph.D., Principal Investigator — George Mason University
Locations (1):
- George Mason University, Fairfax, Virginia, United States

REFERENCES:
- [Derived] Esposito-Smythers C, Hadley W, Curby TW, Brown LK. Randomized pilot trial of a cognitive-behavioral alcohol, self-harm, and HIV prevention program for teens in mental health treatment. Behav Res Ther. 2017 Feb;89:49-56. doi: 10.1016/j.brat.2016.11.005. Epub 2016 Nov 12. PMID 27883927